CLINICAL TRIAL: NCT00794586
Title: A Phase 2, Double-Blind, Multicenter, Randomized, Placebo-Controlled Trial Evaluating Fosfomycin/Tobramycin for Inhalation in Patients With Cystic Fibrosis and Pseudomonas Aeruginosa
Brief Title: Study Evaluating Fosfomycin/Tobramycin for Inhalation in Cystic Fibrosis Patients With Pseudomonas Aeruginosa Lung Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-207-0103
Record Dates: First submitted 2008-11-18; First posted 2008-11-20 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; CF; inhaled antibiotic; antipseudomonal antibiotic; tobramycin; fosfomycin; lung infection; pseudomonal infection; FTI
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FTI 80mg/20mg BID (Experimental): Fosfomycin/Tobramycin combination 80mg/20 mg inhaled twice daily
  Interventions: Drug: FTI, AZLI
- FTI 160mg/40mg BID (Experimental): Fosfomycin/Tobramycin combination 160 mg/40 mg inhaled twice daily
  Interventions: Drug: FTI, AZLI
- Placebo A BID (Placebo Comparator): Placebo A inhaled twice daily
  Interventions: Drug: Placebo, AZLI
- Placebo B BID (Placebo Comparator): Placebo B inhaled twice daily
  Interventions: Drug: Placebo, AZLI

INTERVENTIONS:
Drug: FTI, AZLI — Evaluation of 2 dosage combinations of fosfomycin and tobramycin inhaled twice daily for 28 days following 28 days of inhaled AZLI (Aztreonam Lysine for Inhalation)
  Arms: FTI 160mg/40mg BID; FTI 80mg/20mg BID
Drug: Placebo, AZLI — Volume-matched placebo inhaled twice daily for 28 days following 28 days of AZLI (Aztreonam Lysine for Inhalation).
  Arms: Placebo A BID; Placebo B BID

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 2 dose combinations of fosfomycin/tobramycin for inhalation (FTI), following a 28-day course of Aztreonam for Inhalation (AZLI) in patients with cystic fibrosis and Pseudomonas aeruginosa lung infection.

DETAILED DESCRIPTION:
Gilead is developing a broad spectrum combination antibiotic (FTI) consisting of fosfomycin (an antibiotic with activity against gram-positive and gram-negative bacteria) and tobramycin (an aminoglycoside antibiotic with potent gram-negative activity) for treatment of patients with CF. FTI offers a potential option for treatment of CF lung infections. It is important to note that the concentration of tobramycin in FTI is lower than that of the approved dose of inhaled tobramycin alone, thereby demonstrating the potential of FTI to minimize long-term toxicity from repeated exposure to aminoglycosides like tobramycin. This study will evaluate the safety and efficacy of 2 dose combinations of fosfomycin/tobramycin for inhalation (FTI), following a 28-day course of Aztreonam for Inhalation (AZLI) in patients with cystic fibrosis and Pseudomonas aeruginosa lung infection.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years and older
* Patients with CF as diagnosed by one of the following:

  * Documented sweat chloride greater than or equal to 60 mEq/L by quantitative pilocarpine iontophoresis test, OR
  * Documented sweat sodium greater than or equal to 60 mmol/L, OR
  * Abnormal nasal potential difference, OR
  * Two well-characterized genetic mutations in the CF transmembrane conductance regulator (CFTR) gene, AND
  * Accompanying symptoms characteristic of CF
* Documented presence of PA in an expectorated sputum or throat swab culture at Visit 1 OR documented PA in 2 expectorated sputum or throat swab cultures within 12 months prior to Visit 1; one of the previous PA-positive cultures must be within 3 months prior to Visit 1
* Patients must be able to provide written informed consent prior to any study related procedures
* FEV1 greater than or equal to 25% and less than or equal to 75% predicted at Visit 1
* Ability to perform reproducible pulmonary function tests
* Chest radiograph at Visit 1 without significant acute findings (e.g., infiltrates [lobar or diffuse interstitial], pleural effusion, pneumothorax); or chest radiograph, CT, or MRI obtained within the 90 days prior to Visit 1 without acute findings or significant intercurrent illness; chronic, stable findings (e.g., chronic scarring or atelectasis) are allowed.

Exclusion Criteria:

* Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone a day or 20 mg prednisone every other day
* History of sputum or throat swab culture yielding B. cepacia in the previous 2 years
* Current requirement for daily continuous oxygen supplementation or requirement for more than 2 L/minute at night
* Administration of any investigational drug or device within 28 days of Visit 1 or within 6 half-lives of the investigational drug (whichever is longer)
* Known local or systemic hypersensitivity to monobactam antibiotics
* Known allergies/intolerance to tobramycin or other aminoglycosides
* Known allergies/intolerance to fosfomycin
* Inability to tolerate inhalation of a short acting beta2 agonist
* Changes in or initiation of chronic azithromycin treatment within 14 days prior to Visit 1
* Administration of antipseudomonal antibiotics by inhalation, IV, or oral routes within the 14 days prior to Visit 1
* Changes in antimicrobial, bronchodilator (BD), corticosteroid, hypertonic saline, or dornase alfa medications within 7 days prior to Visit 1
* Changes in physiotherapy technique or schedule within 7 days prior to Visit 1
* History of lung transplantation
* Abnormal renal or hepatic function or serum chemistry at Visit 1, defined as:

  * AST, ALT > 3 times upper limit of normal range (ULN)
  * Creatinine > 1.5 times ULN
* Positive pregnancy test at Visit 1; all women of childbearing potential will be tested
* Female patients of childbearing potential who are lactating or are not (in the opinion of the investigator) practicing an acceptable method of birth control; female patients who utilize hormonal contraceptives as a birth control method must have used the same method for at least 3 months before study dosing
* Any serious or active medical or psychiatric illness, which in the opinion of the investigator, would interfere with patient treatment, assessment, or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Relative change in lung function from baseline at Day 28. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trapnell, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (35):
- United States (35):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Palo Alto, California
  - Denver, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Glenview, Illinois
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Las Vegas, Nevada
  - Albany, New York
  - Buffalo, New York
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Portsmouth, Virginia
  - Richmond, Virginia
  - Tacoma, Washington